CLINICAL TRIAL: NCT01752296
Title: Psychological Concomitants of Morquio Syndrome
Brief Title: Psychological Concomitants of Morquio Syndrome (The MAP Study)
Acronym: MAP
Status: Completed | Type: Observational
Sponsor: Nadia Ali, PhD (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Nadia Ali, PhD, Health Psychologist / Instructor, Emory University
Organization: Emory University (Other)
Other Study IDs: IRB00058524; BioMarin-1 (Other: Other)
Record Dates: First submitted 2012-12-13; First posted 2012-12-19 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Morquio Disease; Mucopolysaccharidosis IV
Keywords: Morquio; Mucopolysaccharidosis IV; Psychological health
MeSH Terms: conditions — Mucopolysaccharidosis IV; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Mucopolysaccharidosis IV, also known as MPS IV or Morquio disease, is a rare autosomal recessive genetic lysosomal storage disorder. Research thus far regarding lysosomal storage diseases (LSDs) in general, including Morquio, has primarily focused on exploring the causes of and finding a treatment for the physical aspects of the various diseases. Less attention has been paid to the psychological or emotional toll of these diseases, whether they are direct symptoms of the diseases themselves or reactions to living with a chronic progressive disease.

It is well established in the health psychology literature, however, that the interaction between our physical health and our psychological health is bidirectional; that is, just as our physical health affects us emotionally (e.g. chronic pain can contribute to depression), so can our psychological health affect us physically (e.g. anxiety can contribute to feelings of chest pain). It is thus critically important to pay attention to the emotional and psychological symptoms associated with all lysosomal storage diseases, including Morquio, and expand our treatment standard of care to include mental health treatment, if necessary.

The first step in understanding and treating psychological conditions in Morquio disease is determining the natural occurrence of psychological symptoms in this population in comparison with non-medical populations. As little has been done in this regard, a pilot study documenting the occurrence rate of psychological issues and overall quality of life in patients with Morquio is the first item in order and will be the focus of this study.

Approximately 20 patients with Morquio disease will be invited to participate, recruited through Emory's Lysosomal Storage Disease Center, as well as through attendance at Morquio support groups and relevant regional, national and/or international meetings. Once consented, patients will be asked to complete three different self-report questionnaires, including the Achenbach System of Empirically Based Assessment (ASEBA) Adult Self-Report (ASR) or Older Adult Self-Report (OASR) questionnaire, the Short Form 36-item Health Questionnaire (SF-36), and the Brief Pain Inventory (BPI). Group aggregate data only will be reported; individual questionnaire content and results will be held confidential, except as in accordance with Georgia law relating to reporting of child or elder abuse, suicidal and/or homicidal intent. Completion of these questionnaires will complete subjects' participation in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Documented clinical diagnosis of MPS IV based on clinical signs and symptoms of MPS IV and documented reduced fibroblast or leukocyte GALNS enzyme activity or genetic testing confirming diagnosis of MPS IV.
2. Patient is at least 18 years old.
3. Patient is not currently receiving enzyme replacement therapy for MPS IV.
4. Patient must provide written, informed consent prior to study participation.

Exclusion Criteria:

1. Previous treatment with ERT
2. Previous hematopoietic stem-cell transplant
3. Patient has a clinically significant disease (with the exception of symptoms of Morquio), including clinically significant immunologic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstances that, in the opinion of the investigator, would confound the effects of Morquio upon study variables

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Morquio Disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
ASEBA Self-Report | At enrollment, as a single-timepoint only
  Self-report questionnaire assessing psychological and adaptive functioning well-being

SECONDARY OUTCOMES:
Brief Pain Inventory | At enrollment, as a single-timepoint only
  Self-report measure of subjective pain levels and interference of pain in daily functioning
SF-36 | At enrollment, as a single-timepoint only
  Brief self-report measure of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ali, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University, Decatur, Georgia, United States